CLINICAL TRIAL: NCT02030210
Title: Quality of Care for STEMI - Patients. a Research to Determine Appropriateness of STEMI Quality Indicators in Belgium, a RAND/UCLA Modified Delphi Study
Brief Title: CP4ACS - Delphi Study to Determine Appropriateness of STEMI Quality Indicators in Belgium
Status: Completed | Type: Observational
Sponsor: European Pathway Association (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Kris Vanhaecht, Study director, European Pathway Association
Other Study IDs: CP4ACS\2013\1
Record Dates: First submitted 2014-01-05; First posted 2014-01-08 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: STEMI; Quality Indicators
Keywords: Quality improvement; STEMI; Belgium
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- cardiologists
- study coordinators
- registred nurses

SUMMARY:
RAND/UCLA modified Delphi study on quality indicators for STEMI to determine the appropriateness of quality indicators retrieved from literature and guideline review. We aim to engage 20 cardiologists and 20 nurses with relevant experience in the care for STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* cardiologist or cardio nurse with relevant experience in the care for STEMI patients

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We aim to engage 20 cardiologists and 20 cardio nurses, all experienced in the care for STEMI patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
validated quality indicators for STEMI care in belgium (both on patient and on hospital level) | 2 months
  33 experts in cardioloy, cardio nursing and quality rated quality indicators for STEMI care in belgian hospitals on a 9 point Likert Scale. All indicators with a median score between 7 and 9 were discussed in an expert panel. The expert panel selected validated quality inidicators for STEMI care.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Vanhaecht, dr, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams Brabant, Belgium